CLINICAL TRIAL: NCT06409299
Title: Enhancing Lung Health in Kids With Structural Lung Damage and Malformations: a Randomized Controlled Trial on Azithromycin (AZI) for Airway Infection Prevention
Brief Title: Enhancing Lung Health in Kids With Structural Lung Damage and Malformations: Azithromycin (AZI) for Airway Infection Prevention
Acronym: TRALULALA-AZI
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Marika Nathalie Schmidt, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: p-2024-15966
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Tracheomalacia; Bronchopulmonary Dysplasia (BPD); Vascular Ring; Cystic Lung Disease; Bronchiectasis; Chronic Atelectasis
MeSH Terms: conditions — Tracheomalacia; Bronchopulmonary Dysplasia; Vascular Ring; Cystic Disease Of Lung; Bronchiectasis | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: The study comprises a multicenter, parallel-group, double-blind, randomized placebo-controlled clinical trial (RCT) with a single intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin Oral Suspension 40 mg/ml (Active Comparator)
  Interventions: Drug: Azithromycin 40 MG/ML
- Placebo Oral suspension (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Azithromycin 40 MG/ML — Maintenance Antibiotic treatment
  Arms: Azithromycin Oral Suspension 40 mg/ml
Other: Placebo — Placebo
  Arms: Placebo Oral suspension

SUMMARY:
Children with lung and airway malformations or early structural lung damage face significant challenges, often leading to recurrent respiratory infections, hospitalizations, and decreased quality of life. Despite various interventions, effective strategies are urgently needed.

The link between these conditions and persistent bacterial bronchitis remains unclear, possibly due to compromised airways and reduced mucociliary clearance. Although antibiotics can alleviate symptoms, relapse is common.

Experts often prescribe prophylactic azithromycin, despite limited evidence of its benefits. Azithromycin shows promise due to its anti-inflammatory and immunomodulatory effects but lacks thorough evaluation in this population.

To address this gap, we propose a double-blind, randomized controlled trial to assess azithromycin's effectiveness and safety in preventing respiratory infections in children with these conditions. This research aims to inform clinical practice and improve the health of affected children and their families.

ELIGIBILITY:
Inclusion Criteria:

1. CT and bronchoscopy verified and structural lung damage or congenital lung and airway malformations
2. Outpatient affiliation with one of the three highly specialized pediatric pulmonology centers.
3. At risk of or already documented respiratory infections requiring antibiotics.
4. Age between 0-72 months at inclusion.

Exclusion Criteria:

1. Asthmatic challenges: Patients without any of the conditions mentioned in table 1 repeatedly experiencing asthmatic problems are not eligible for this study.
2. Cystic fibrosis (CF) or primary ciliary dyskinesia (PCD): Patients with a CF or PCD diagnosis will be excluded.
3. Impaired liver function: Children with an alanine transaminase (ALAT) twice or more the upper limits of normal will be excluded.
4. Impaired kidney function: Children with a serum creatinine higher than the upper limit of normal for age will be excluded.
5. Neurological or psychiatric disorders
6. Prolonged QT interval: Patients with either congenital or acquired prolonged QT interval will be excluded.
7. Heart disease: Patients with clinically relevant bradycardia, cardiac arrhythmia or severe heart failure are not eligible for this study.
8. Allergy to macrolide antibiotics: documented allergy to macrolide antibiotics (extremely rare) will result in exclusion from the study.

Ages: 0 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of exacerbations | 6 months
  Number of exacerbations where systemic antibiotics is needed within the study period

SECONDARY OUTCOMES:
Severity of exacerbations | 6 months
  Duration of exacerbations, hospitalizations and durations of hospitalizations

OTHER OUTCOMES:
Lung function measures | 1 year
  Impulse oscillometry (IOS) measurement pre- and post drug administrations
Quality of Life | 1 year
  Questionaire on a Likert scale 0-5. Using PedsQL(TM).

IPD SHARING:
Plan to Share IPD: Undecided